CLINICAL TRIAL: NCT05235178
Title: The Effect of the CytoSorb® Filter to Remove Anticoagulants From the Circulation During Emergency Surgery for Aortic Dissection
Acronym: Citron
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Johannes Lagethon Bjørnstad, Consultant Surgeon and Associate Professor, Oslo University Hospital
Other Study IDs: 20/27731
Record Dates: First submitted 2022-01-05; First posted 2022-02-11 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Aortic Dissection; Factor X Inhibition
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Due to catastrophic bleeding events in patients who are anticoagulated with FXa inhibitors undergoing emergency surgery on the proximal aorta and lack of antidote (not available in Norway and most likely not compatible with heparin), the department has decided to use hemadsorber in these cases.

SUMMARY:
The direct oral anticoagulants (DOACs) and particularly the FXa inhibitors are a concern in patients presenting with type A aortic dissection as this may contribute to severe bleeding complications. The antidote andexanet alfa (Ondexxya®) can interact with the heparin- anti-thrombin III (ATIII) complex which may neutralize the anticoagulant effect of heparin and the use of andexanet alfa before surgery necessitating heparin-anticoagulation has been reported to cause unresponsiveness to heparin. The investigators have preliminary in-vitro data demonstrating the ability to remove apixaban from reconstituted blod by hemadsorption and are now analyzing if aFXa inhibitor levels may be reduced by hemadsorption in the clinical setting analyzing this in patients using FXa inhibitors being operated acutely for type A aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Indication for urgent surgery for proximal aortic disease
* Treatment with FXa inhibitor for more than 2 weeks
* Measured concentration of FXa inhibitor in therapeutic range (>50 ng/mL) at the time of admission.
* Intraoperative use of Cytosorb® hemadsorber.

Exclusion Criteria:

• Low FXa inhibitor concentration (<50 ng/mL) at the time of admission

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are anticoagulated with FXa inhibitors beeing operated acutely for acute proximal aortic disease with the use of Cytosorb® hemadsorber intraoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Change in apixaban concentration after 60 minutes of hemadsorption | 60 minutes
  Apixaban concentration will be analysed by ultraperformance liquid chromatography mass spectrometry (UPLC-MS) from blood samples at different time-points (0, 5, 10, 30, 60, 120 minutes) during hemadsorption.

SECONDARY OUTCOMES:
Change in apixaban concentration during hemadsorption | 5-120 minutes
  Apixaban concentration will be analysed by ultraperformance liquid chromatography mass spectrometry (UPLC-MS) from blood samples at different time-points (0, 5, 10, 30, 60, 120 minutes) during hemadsorption.
Apixaban concentration follwing hemadsorption | 24 hours
  Apixaban concentration will be analysed by ultraperformance liquid chromatography mass spectrometry (UPLC-MS) from blood samples 24 hours after hemadsorption.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway